CLINICAL TRIAL: NCT03194256
Title: Effects of Very Low Nicotine Content Cigarettes and E-cigarette Characteristics on Smoking in Adolescents
Brief Title: Evaluating New Nicotine Standards for Cigarettes - Project 3
Acronym: CENIC2-P3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Wake Forest University (Other); University of Minnesota (Other); National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1705001771; U54DA031659 (NIH)
Record Dates: First submitted 2017-06-07; First posted 2017-06-21 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Smoking, Cigarette; Electronic Cigarettes
Keywords: Smoking; Cigarettes; E-Cigarettes
MeSH Terms: conditions — Cigarette Smoking; Vaping; Smoking

STUDY DESIGN:
Intervention Model Description: Mixed between subjects and within-subjects design. Random assignment to the between subjects factor (nicotine content in cigarettes), within-subjects manipulation of nicotine concentration and flavors in e-liquid in the electronic cigarettes
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blind to the nicotine content of their assigned study cigarette and the nicotine dose of the e-liquid in the study vaping device. Investigators, research staff, and biostatisticians will also be blind to the conditions. E-liquid flavors will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Nicotine Content Cigarettes (Active Comparator): Spectrum Research Cigarettes: 15.8 mg nicotine/g tobacco, 9 mg of tar
  Interventions: Behavioral: Spectrum Research Cigarettes
- Very Low Nicotine Content Cigarettes (Experimental): Spectrum Research Cigarettes: 0.4 mg nicotine/g tobacco, 9 mg of tar
  Interventions: Behavioral: Spectrum Research Cigarettes

INTERVENTIONS:
Behavioral: Spectrum Research Cigarettes — Participants will be assigned to either normal nicotine content cigarettes or very low nicotine content cigarettes.

SUMMARY:
This study is designed to examine how the nicotine content of cigarettes and the nicotine concentration and flavors in e-liquids influence responses to and use of these products in adolescent smokers. Participants will complete a total of six sessions (an in-person screening/baseline session and five lab sessions.

DETAILED DESCRIPTION:
Adolescence is a critical developmental period for tobacco initiation and progression to regular use and dependence. The Food and Drug Administration (FDA) has the authority to establish standards for tobacco products for the protection of public health, including the authority to mandate a reduction in the nicotine content of all cigarettes to minimally addictive levels. Numerous studies have found that adult smokers who are switched to very low nicotine content (VLNC) cigarettes experience reductions in smoking rates, nicotine intake, nicotine dependence and abstinence-induced craving relative to those who use normal nicotine content (NNC) cigarettes. However, studies of VLNC cigarettes in adolescent smokers are limited and more information is needed to inform potential product standards. Furthermore, use of electronic nicotine delivery systems (ENDS), e-cigarettes or vaping devices, has increased dramatically in adolescents. Therefore, effects of VLNC cigarettes on smoking in youth should be examined in the context of vaping device availability. This study is designed to examine how the nicotine content of cigarettes and the nicotine concentration and flavors in e-liquids influence responses to these products in adolescents.

Participants will complete an in-person baseline session in which eligibility criteria are confirmed and background questionnaires are completed. Next, participants will complete five in-person lab sessions in which NNC or VLNC cigarettes are available (based on random assignment). During the first lab session, participants will test the assigned research cigarettes when no alternative product is available. During each of the four remaining lab sessions, smokers' responses to the assigned research cigarettes will be compared to their responses to a vaping device with the following characteristics: 1) no nicotine, tobacco flavor; 2) no nicotine, non-tobacco flavor; 3) moderate nicotine concentration, tobacco flavor; or 4) moderate nicotine concentration, non-tobacco flavor. In each session, after sampling and rating the subjective effects of the products available during that session, participants will make a series of 10 choices. Choices will be for either 2 puffs of the research cigarette, 2 puffs of the vaping device, or abstinence from puffing.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 15-20
2. Adolescents who report current daily or near daily cigarette smoking for at least 3 months
3. Must have used an electronic nicotine device on a minimum of two lifetime occasions.
4. Breath Carbon Monoxide (CO) levels > 5 ppm (if < 5 ppm, then cotinine assay via NicAlert Strip = > 3)
5. Speak, comprehend, and read English well enough to complete study procedures

Exclusion Criteria:

1. Unwilling to use research cigarettes or ENDS as part of the study
2. Intention to quit smoking in the next 30 days
3. Using tobacco products (other than ENDS or roll-your-own tobacco) > 15 days in the past 30 days.
4. Any medical or psychiatric condition in which participation is likely to post a significant threat to health or for which the condition could interfere with the ability of the participant to fully participants (as determined by the LMP)
5. Self-reported illicit use of any drug except marijuana > 10 days in the past 30 days
6. Binge drinking alcohol (>10 days in the past 30 days, >4/5 drinks in a 2-hour period (female/male))
7. Pregnant or breastfeeding
8. CO reading > 80 ppm
9. Systolic BP outside the range of 90-159, diastolic BP outside the range of 50-99, or heart rate outside the range of 45-104. Participants failing for any of these criteria will be allowed to re-screen once per criterion.
10. Indicating Yes on Questions 4-6 on the MINI with a suicide attempt in the past 2 years (if within the past 2-10 years, LMP approval required).
11. Having participated in another research study during the past year in which they were switched to reduced nicotine cigarettes for longer than one week.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Colby, PhD, Principal Investigator — Brown University; Jennifer Tidey, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Intend to share findings from this research through publications and presentations. Institutions and individuals wishing to access any resources or data must contact the Principal Investigator (Hatsukami). Data will be available in two formats. One will be a summary of the data, with graphs and tables, posted as pdf files and as raw individual-level data for analysis. Data generated by this grant will be made to outside investigators, according to NIH Guidance. When data are shared, there will be no limits placed on how the data will be used. Users will agree, however, that the recipient must not transfer the data to other users and that the data are only to be used for research purposes. A record of transfer of data and a copy of the dataset that was distributed will be kept by Brown University.
Time Frame: Data will not be available until primary and secondary papers are accepted for publication.
Access Criteria: Persons requesting data must do so in writing, identifying their affiliation and how the data will be used. Upon review, access will be determined.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Started | 41 | 39
Laboratory Session 2 | 41 | 36
Laboratory Session 3 | 40 | 33
Laboratory Session 4 | 39 | 33
Completed | 38 | 32
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Population: Participants who were randomized at Lab Session 1
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.9 (.7) | 18.7 (0.8) | 18.8 (0.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 24 | 22 | 46
  Transgender male to female | 1 | 1 | 2
  Transgender female to male | 0 | 0 | 0
  Genderqueer/gender non-conforming | 2 | 0 | 2
  Different identity | 0 | 1 | 1
  Prefer not to answer | 1 | 0 | 1
  Unknown | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 32 | 34 | 66
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 27 | 24 | 51
  More than one race | 8 | 5 | 13
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 80
Average Cigarettes Per Day [Mean (Standard Deviation); unit: Cigarettes smoked per day] | 5.8 (5.6) | 4.7 (3.6) | 5.3 (4.7)
Fagerstom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — The Fagerstrom Test for Nicotine Dependence scale total score ranges from 0-10, with higher scores indicating greater dependence.
  units on a scale | 2.6 (2.2) | 2.2 (1.7) | 2.4 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Cigarette Puffs Taken (0 to 20)
Description: The number of cigarette puffs selected during a 30 minute choice procedure when no vaping device was available
Time Frame: 30-minute preference task
Population: Laboratory session 1
Measure: Mean (Standard Deviation); unit: Puffs chosen
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 41 | 39
Puffs chosen | 12.1 (5.0) | 10.8 (5.3)

2. Primary Outcome: Number of Cigarette Puffs Taken (0 to 20) When the Available Vaping Device Has 3mg/ml of Nicotine and Was Available in Tobacco Flavor
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device has 3mg/ml of nicotine and was available in tobacco flavor
Time Frame: 30-minute preference task
Population: Counterbalance laboratory sessions 2-5
Measure: Mean (Standard Deviation); unit: Puffs chosen
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 33
Puffs chosen | 8.9 (5.6) | 5.2 (5.4)

3. Primary Outcome: Number of Cigarette Puffs Taken (0 to 20) When the Available Vaping Device Has 3mg/ml of Nicotine and Was Available in Non-tobacco Flavors
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device has 3mg/ml of nicotine and was available in non-tobacco flavors
Time Frame: 30-minute preference task
Population: Counterbalanced laboratory sessions 2-5
Measure: Mean (Standard Deviation); unit: Puffs chosen
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 40 | 34
Puffs chosen | 8.0 (5.0) | 4.6 (4.3)

4. Primary Outcome: Number of Cigarette Puffs Taken (0 to 20) When the Available Vaping Device Has 18mg/ml of Nicotine and Was Available in Tobacco Flavor
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device has 18mg/ml of nicotine and was available in tobacco flavor
Time Frame: 30-minute preference task
Population: Counterbalanced laboratory sessions 2-5
Measure: Mean (Standard Deviation); unit: Puffs chosen
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 33
Puffs chosen | 9.4 (5.4) | 4.7 (5.1)

5. Primary Outcome: Number of Cigarette Puffs Taken (0 to 20) When the Available Vaping Device Has 18mg/ml of Nicotine and Was Available in Non-tobacco Flavors
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device has 18mg/ml of nicotine and was available in non-tobacco flavors
Time Frame: 30-minute preference task
Population: Counterbalanced laboratory sessions 2-5
Measure: Mean (Standard Deviation); unit: Puffs chosen
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 34
Puffs chosen | 8.6 (5.4) | 4.5 (4.2)

6. Secondary Outcome: Number of E-cig Puffs Taken (0 to 20) When the Available Vaping Device Contained 3mg/ml Nicotine and Was Available in Tobacco Flavor
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device contained 3mg/ml nicotine and was available in tobacco flavor
Time Frame: 30-minute preference task session
Measure: Mean (Standard Deviation); unit: vape puffs
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 33
vape puffs | 6.6 (5.0) | 10.5 (6.1)

7. Secondary Outcome: Number of E-cig Puffs Taken (0 to 20) When the Available Vaping Device Contained 3mg/ml Nicotine and Was Available in Non-tobacco Flavors
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device contained 3mg/ml nicotine and was available in non-tobacco flavors
Time Frame: 30-minute preference task session
Population: Counterbalance laboratory session 205
Measure: Mean (Standard Deviation); unit: vape puffs
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 40 | 34
vape puffs | 7.2 (4.6) | 11.0 (6.0)

8. Secondary Outcome: Number of E-cig Puffs Taken (0 to 20) When the Available Vaping Device Contained 18mg/ml Nicotine and Was Available in Tobacco Flavor
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device contained 18mg/ml nicotine and was available in tobacco flavor
Time Frame: 30-minute preference task session
Measure: Mean (Standard Deviation); unit: vape puffs
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 33
vape puffs | 4.3 (4.3) | 8.2 (6.6)

9. Secondary Outcome: Number of E-cig Puffs Taken (0 to 20) When the Available Vaping Device Contained 18mg/ml Nicotine and Was Available in Non-tobacco Flavors
Description: The number of cigarette puffs selected during a 30 minute choice procedure when the available vaping device contained 18mg/ml nicotine and was available in non-tobacco flavors
Time Frame: 30-minute preference task session
Measure: Mean (Standard Deviation); unit: vape puffs
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 34
vape puffs | 5.2 (5.0) | 11.0 (5.6)

10. Secondary Outcome: Carbon Monoxide Change From pre-to the Post-choice Task When no Vaping Device Was Available
Description: Post-choice CO minus pre-choice CO at session 1 in which no vaping device was available
Time Frame: 30-minute preference task
Population: Laboratory session 1
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 41 | 39
parts per million | 5.9 (4.3) | 6.7 (4.5)

11. Other Pre Specified Outcome: Number of Choices for Cigarette Puffs
Description: 0 to 10
Time Frame: 30-minute preference task at each of the 5 laboratory sessions
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Choices for E-cig Puffs
Description: 0 to 10
Time Frame: 30-minute preference task at each of the 5 laboratory sessions
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Number of Choices to Abstain From Puffing
Description: 0 to 10
Time Frame: 30-minute preference task at each of the 5 laboratory sessions
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Drop-out Rate
Description: Measures of compliance
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Minnesota Nicotine Withdrawal Scale (MNWS)
Description: Measures withdrawal symptoms
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Questionnaire of Smoking Urges (QSU)
Description: Measures craving
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Positive and Negative Affect Scale (PANAS)
Description: Measures positive and negative affect
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Cigarette Evaluation Scale (CES)
Description: Measures subjective responses cigarettes
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Cigarette Purchase Task
Description: Measures demand for cigarettes across a range of prices
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Perceived Health Risk Scale
Description: Measures perceived risk of cigarettes
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Heart Rate
Description: Measures of cardiovascular function
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Blood Pressure
Description: Measures of cardiovascular function
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Total Nicotine Equivalents (TNE)
Description: Biomarkers
Time Frame: Baseline; Week 1
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Nicotine Metabolite Ratio (NMR)
Description: Biomarkers
Time Frame: Baseline; Week 1
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Cotinine
Description: Biomarkers: measures a metabolite of nicotine
Time Frame: Baseline; Week 1
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Carbon Monoxide (CO)
Description: Biomarkers: measures expired alveolar carbon monoxide level
Time Frame: Baseline-Lab Session 5; 2-8 weeks; average 3-4 weeks
Reporting Status: Not Posted

27. Secondary Outcome: Carbon Monoxide Change From pre-to the Post-choice Task When the Available Vaping Device Contained 3mg/ml Nicotine and Was Available in Tobacco Flavor
Description: Post-choice CO minus pre-choice CO when the available vaping device contained 3mg/ml nicotine and was available in tobacco flavor
Time Frame: 30-minute preference task
Population: Laboratory session 1
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 33
parts per million | 4.4 (3.2) | 3.8 (3.2)

28. Secondary Outcome: Carbon Monoxide Change From pre-to the Post-choice Taskwhen the Available Vaping Device Contained 3mg/ml Nicotine and Was Available in Non-tobacco Flavors
Description: Post-choice CO minus pre-choice CO when the available vaping device contained 3mg/ml nicotine and was available in non-tobacco flavors
Time Frame: 30-minute preference task
Population: Counterbalanced laboratory sessions 2-5
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 40 | 34
parts per million | 3.9 (3.6) | 3.6 (2.9)

29. Secondary Outcome: Carbon Monoxide Change From pre-to the Post-choice Task When the Available Vaping Device Contained 18mg/ml Nicotine and Was Available in Tobacco Flavor
Description: Post-choice CO minus pre-choice CO when the available vaping device contained 18mg/ml nicotine and was available in tobacco flavor
Time Frame: 30-minute preference task
Population: Counterbalanced laboratory sessions 2-5
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 33
parts per million | 4.3 (3.4) | 2.7 (2.1)

30. Secondary Outcome: Carbon Monoxide Change From pre-to the Post-choice Task When the Available Vaping Device Contained 18mg/ml Nicotine and Was Available in Non-tobacco Flavors
Description: Post-choice CO minus pre-choice CO when the available vaping device contained 18mg/ml nicotine and was available in non-tobacco flavors
Time Frame: 30-minute preference task
Population: Counterbalanced laboratory sessions 2-5
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
Number analyzed (Participants) | 39 | 34
parts per million | 4.0 (2.4) | 3.3 (3.5)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each of 5 laboratory sessions, which occurred 2-7 days apart. The shortest assessment time (i.e., from the first to the last session) was 12 days; the longest was 40 days. At the 30-day follow-up call, any adverse events that remained open (i.e., were still ongoing) were assessed; no new adverse events were assessed for at the 30-day follow-up call.
Description: SAEs were defined per clinicaltrials.gov definitions. Other (Not Including Serious) Adverse Events were defined as AEs classified as 'severe' by the medical monitor.
Arm/Group | Normal Nicotine Content Cigarettes | Very Low Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT03194256/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT03194256/ICF_001.pdf